# Study protocol cover page

Official study title: Multicenter registry to study the characteristic and outcomes of Jordanian Heart Failure patients

The Jordanian Heart Failure Registry (JoHFR)

NCT04829591

The actual document date and approval date 30/3/2021

The updated document date 17/4/2021

# A Multicenter Registry to Study the Characteristics and Outcomes of Jordanian Heart Failure Patients.

The Jordanian Heart Failure Registry (JoHFR)

ClinicalTrials.gov Identifier: NCT04829591

### (Study protocol)

Principal investigator and study chair: Hadi Abu-Hantash, MD, MSc, FACC, FSCAI.

Principal investigator: Mahmoud Izraiq, MD.

# **Brief Summary**

Heart Failure research registry is a collection of computerized information about individuals with heart failure. The database in this registry is obtained from several Jordanian medical centers which will represent an extremely valuable resource for epidemiological research on heart failure patients.

## **Detailed Description:**

Understanding the cause of Heart Failure (HF) and how the body will respond to it, is critical for an effective treatment. HF is a global problem with significant morbidity and mortality, despite improved understanding of the pathophysiology and a growing range of therapeutic options. Jordanian Heart Failure Registry (JoHFR) will be the first research project of heart failure prevalence in Jordan. It is undertaken by primary healthcare professionals with main aim to improve knowledge about the care of patients with HF. The investigators responsible for conducting this research are physicians and their teams who deal with heart failure patients in their outpatient and inpatient clinic centers including the public and private medical sectors in Jordans' medical community. Standards in the Hashemite kingdom of Jordan complies with the recognized good guideline directed medical practices internationally.

#### **Objectives of the registry:**

Up to date, there is still a lack of reliable pathology data that summarizes patient cases with heart failure disease. This research aims to fill this gap and provide the local and international medical communities with this important set of comparative data in order to determine our current situation in regards to screening, management, and follow up of patients. This will have a direct impact on improving Heart Failure patient outcomes by directing our focus on strengths and weaknesses in our management in this ongoing high morbidity and mortality syndrome. Furthermore, this registry will focus on describing the diagnostic and therapeutic approaches undertaken by cardiologists in their care of patients with HF in order to improve future management

of patients with high HF risks. The prevalence of the clinical profiles of patients with acute and chronic HF will also be evaluated.

### Study design and methodology:

- This registry consists of multiple variables including demographics, concomitant diseases, diagnostic procedures, hemodynamics, laboratory data, and medications used, discharge information and instructions. The patient information is detailed in the attached questionnaire (appindex1) which will be filled by participating who will record details of their HF patients and transfer these data for documentation.
- This study aims to include sufficient number of patients with Heart Failure and is expected to last for extended time until the study sample is completed by participating healthcare professionals. The data collected at 12 months will be the basis of the initial statistics, upon which the trial duration will be determined.
- The principal research coordinator and his team will train personnel of the participating units on how to register patients and how to use the registry.
- Patient safety, security and confidentiality will be retained at all times during the course of the study and thereafter.
- Follow up after one year should include data on morbidity (including Heart failure hospitalization) and mortality with detailed information on medications, quality of life, and functional capacity. The study will comply with the ethics of research and (IRB) institutional review board approvals and any other required official organizational requirements.

### Inclusion and exclusion criteria:

- Inclusion criteria:
  - 1. Patients who are 18 years or older with Heart Failure diagnosis as defined by internationally recognized guidelines.
  - 2. Current residents of the Hashemite Kingdom of Jordan.
- Exclusion criteria:
  - 1. Patients who refuse or unable to sign a consent form.
  - 2. Patient inability to follow up with provider

#### **Statistical analysis:**

Data will be pooled and descriptive and comparative statistical tests will be used to categorize the patients based on the disease sub-typing and management quality and to find the prevalence of heart failure disease different types, classes and stages amongst Jordanians. Furthermore, comparative analysis will be performed to test the efficiency, accuracy, and the quality of medical practice in Jordan. Statistical analysis will be done using SPSS V21.

See appindex1 below.

| ex |
|----|

| Chronic HF ☐ Acute HF ☐ | Patient Initials/Site number: |
|---|---|
| DOB: / / (MM/DD/YYYY) Gender: M F Admission date/ Office visit / / : | |
| Discharge Date/Time / / : | |

| | Medical History (Select all that apply): | |
|---|---|---|
| □ H/O ASCVD | □ Implanted devices | □ Notes : |
| □ H/O Arrhythmias | □ History of structural heart disease | |
| | □ Other relevant medical history | |
| □ ASCVD risk factor: | | |
| <b>♦♦</b> DM | | |
| �� HTN | | |
| <b>♦♦</b> Smoking | | |
| ♦♦ Alcohol<br>Abuse | | |
| <b>♦♦</b> Dyslipidemia | | |
| <b>♦♦</b> Obesity | | |
| Positive family history of premature ASCVD | | |
| ♦♦ CKD | | |
| Others. | | |
| | Heart Failure History | |
| Etiology: | □ Ischemic/CAD | □ Non-Ischemic |
| Check if history of : | | □ Hypertensive |
| | | □ Alcohol/Other Drug |
| | | □ Chemotherapy |
| | | □ Viral |
| | | □ Postpartum |
| | | □ Familial |
| | | □ Other Etiology |
| | | □ Unknown/Idiopathic |

| Known history of HF prior to this admission? | o Yes | | O No |
|---|---|---|---|
| # of hospital admissions in past 6 mo./office visit for HF: | 0 | 2 | o Unknown |
| | <u> </u> | >2 | |
| 1 | | | |
| 1 | Medications Used Prior to | Admission: [Select all that a | pply] |

| □ Patient on no meds prior to admission □ ACE Inhibitor □ Aldosterone Antagonist □ Angiotensin receptor blocker (ARB) □ Angiotensin Receptor Neprilysin Inhibitor (ARNI) □ Antiarrhythmic □ Aspirin □ Antiplatelet agent (excluding aspirin) | □ Anticoagulation Therapy | □ Beta-Blocker( metoprolol, propranolol, bisoprolol, atenolol, acebutelol, nebivelol, nadolol) □ Ca channel blocker( amlodipine, nefidipine, nicardipine, verapamil, diltiazem) □ Digoxin □ Diuretic □ Thiazide/Thiazide like( chlorothalidone, hydrochlorothiazide, indapamide, metolazone) □ Loop( bumetanide, furosemide, torsemide) □ Hydralazine □ Ivabradine □ Lipid lowering agent (Any) □ Statin( rosuvastatin, atorvastatin, simvastatin, fluvastatin, pravastatin) □ Other Lipid lowering agent □ Nitrate( nitroglycerin, nitroprusside, isosorbide) □ Other |
|---|---|---|
| Symptoms (Closest to Admission) Select all that apply | ☐ Dyspnea ☐ PND NYHA class ☐ Fatigue ( , , , V) ☐ Chest pain ☐ Orthopnea | ☐ Palpitations |

| Vital signs | <b>Height ��</b> cm |
|-------------|---------------------|

| Weight BMI �� Kgs. |
|--------------------|

| Heart Rate | Heart Rate bpm | ☐ Reg | |
|---|---|---|---|
| Examination<br>(Closest to | JVP: O Yes | o No | |
| Admission/Office visit) | Rales: O Yes | o No | |
| | Lower Extremity O Yes Edema | o No | |
| Lipids | TC: LDL: HDL: _ mg/dL mg/dL mg/dL | TG:<br>mg/dL | □ Lipids Not<br>Available |
| Labs Closest to Admission)/ office visit | Na | o mg/dL | ☐<br>Unavailabl e |
| | BNP | o ng/L | ☐<br>Unavailabl e |
| | К | o mg/dL | □<br>Unavailabl e |
| | Hb | o g/dL | □<br>Unavailabl e |
| | Albumin | o g/dL | ☐<br>Unavailabl e |
| | NT-proBNP | o ng/L | ☐<br>Unavailabl e |
| | SCr | o mg/dL | ☐<br>Unavailabl e |

| eGFR | o ml/min/ □ MDRD<br>1.73m² |
|-----------------------------------------------|------------------------------|
| BUN | ○ mg/dL □ Unavailabl e |
| Troponin (Peak) ng/L �� T quantitative / Hs | Normal Unavailabl e Abnormal |
| Ferritin<br>ng/mL<br>Transferrin saturation | |
| HbA1C % | Unavailable |
| Fasting Blood<br>Glucose | Unavailable |
| (mg/dL) EKG QRS | Unavailable |
| Duration (ms) | |
| EKG QRS | <b>♦♦</b> Paced |
| Normal RBB Morphology B LBBB NS IVCD | �� Unavailable |
| Procedures | |

| | ☐ No Procedures | ☐ Atrial Fibrillation Ablation or Surgery |
|---|---|---|
| | ☐ Cardiac Cath/Coronary Angiography | □ Cardiac Valve Surgery |
| | ☐ Coronary Artery Bypass Graft | □ Cardioversion |
| | ☐ CRT-P (cardiac | ☐ CRT-D (cardiac resynchronization therapy |
| | resynchronizationtherapy pacing only) | with ICD ☐ Intra-aortic Balloon Pump |
| ☐ Dialysis or Ultrafiltration ☐ ICD only | | ☐ Left Ventricular Assist Device |
| | · | □ Pacemaker |
| | <ul><li>□ Mechanical Ventilation</li><li>□ PCI</li></ul> | |
| | ☐ Right Cardiac Catheterization | |

| EF | - By Echo - By other means % | Obtained: | <ul><li>♦♦ This Admission</li><li>♦♦ Within the last year</li><li>♦♦ &gt; 1 year ago</li></ul> |
|---|---|---|---|
| Added Oral Medications during hospitalization Select all that apply | □ None □ ARNI □ ARB | ☐ Aldosterone Antagonist ☐ Hydralazine Nitrate | □ ACE Inhibitor □ Beta Blocker |
| Parenteral Therapies<br>during hospitalization<br>Select all that apply | □ None □ Dopamine □ Iron □ Milrinone | <ul><li>□ Nitroglycerine</li><li>□ Other IV</li><li>Vasodilator</li></ul> | <ul> <li>□ Dobutamine</li> <li>□ Loop Diuretics</li> <li>□ Intermittent Bolus</li> <li>□ Continuous Infusion</li> </ul> |

| Was the patient | Yes No | Not Documented |
|------------------------------------------|--------|----------------|
| ambulating at the end of hospital day 2? | | |

| Was DVT prophylaxis initiated by the end of hospital day 2? | Yes | s No | Contrain | dicated |
|---|---|---|---|---|
| If yes, | | onated heparin (LDUH)<br>ar weight heparin | □ Direc | ctor Xa Inhibitor t thrombin inhibitor mittent pneumatic pression devices (IPC) |
| Discharge Date/Time / / : | | | ☐ MM | I/DD/YYYY only |
| Primary Cause of Death | o Cardiovascula | r o Non-Cardiovascular | o Unkn | own |
| If Cardiovascular: | <ul><li>Acute Coronary</li><li>Syndrome</li></ul> | <ul><li>Worsening</li><li>Heart Failure</li></ul> | Suc | dden Death<br>er |
| When is the earliest documents measures only? | ation of comfort | Day 0 or 1 Day 2 or after | | ing unclear<br>Documented |
| Symptoms (closest to discharge) | <ul><li>Worse</li><li>Unchanged</li></ul> | Better, Symptomatic Better, Asymptomatic | Una | able to determine |
| Vital Signs (closest to Discharge) | Weight ��Kgs. | | ☐ Not Documented | |
| | Heart Rate Bpm regu | lar Irregular | □ N | ot Documented |
| | BP-Supine _ / _ mmHg | g (systolic/diastolic) | □ N | ot Documented |
| | Respiratory Rate breat | hs per minute | | |
| Exam (Closest to Discharge) | JVP: o Y | ∕es ○ No | O<br>Unknow<br>n | |
| | Rales: O Yes | | o N | lo |

| | Lower Extremity • Yes | | o <b>No</b> | |
|---|---|---|---|---|
| | Edema | | | |
| Labs (Closest to Discharge) | Na | o mg/dl | L 🔲 Unav | ailable |
| | BNP | o mg/dl | L 🔲 Unav | ailable |
| | SCr | o mg/dL ☐ Unavailable | | |
| | BUN | o mg/dL ☐ Unavailable | | |
| | NT-BNP (pg/mL) | | Not Document | ed |
| | κο mEq/L | o mmol/ | /L o mg/dL | |
| | eGFR •• MI/min/ 1.73m² | | □ N | MDRD |
| | | ·! | | |
| | Angiotensin Converting Enzyme Inhibitor (ACEI) | | | |
| Prescribed? | ∘ Yes ∘ No | | Frequency: | |
| If Yes, | Medication: Dosage: | | | |
| Beta-Blocker | | | | |
| Name: | Dose: | | | |
| Aldosterone Antagonist | | | | |
| Medication: Dosage: Frequency: | | | | |
| Anti-hyperglycemic Medications: | | | | |
| Name: | Dose: | | | |
| Lipid Lowering Medication(s): | | | | |
| Name: | Dose: | | | |
| | Hydralazine Nitrate | | | |

| Name: | Dose: | | |
|---|---|---|---|
| | Other Medications at D | Discharge | • |
| ☐ Antiarrhythmic ☐ Amiodarone ☐ Sotalol ☐ Other | ☐ Ca Channel Blocker ☐ Digoxin ☐ Diuretic ☐ Loop ☐ Diuretic ☐ Thiazide ☐ Diuretic | □ Nitrate □ Ranolazine □ Other Anti-Hypertens □ Other | sive |
| | Angietaneia Decenter Di | ocker (ADD) | |
| | Angiotensin Receptor Blo | ocker (ARB) | |
| Name: | Dose: | | |
| | Angiotensin Receptor Neprilysi | n Inhibitor (ARNI) | |
| Name: | Dose: | | |
| | Acetylsalicylic acid | (ASA) | |
| Name: | Dose: | | |
| | Anticoagulation Th | erapy | |
| Prescribed? | Yes No | | Dosage |
| If Yes, | Class: | ☐ Other | |
| | ☐ Warfarin | | |
| | | • | |
| | □ DOAC | | |
| | Clopidogrel | <u> </u> | |
| Prescribed? | ∘ Yes∘ No | | |

| If Yes, | Dosage: Frequency: | | |
|---|---|---|---|
| | Other Antiplatelet(s) | • | |
| Name: | dose: | | |
| Activity | ○ Yes ○ No Diet (Salt restricted) | o Yes | o No |
| Follow-up | ○ Yes ○ No Medications | o Yes | o No |
| Symptoms Worsening | ○ Yes ○ No Weight Monitoring | o Yes | o No |
| Follow-up Visit Scheduled | <ul><li>Yes </li><li>No Date/Time of first follow up visit:</li></ul> | //: | |
| Location of first follow-up visi | Telehealth Not Documented | | |
| | | • | • |
| Medical or Patient Reason for appointment being scheduled | ∘ Yes | o No | |
| | Follow up visits form: | | |
| Scheduled at: | 3 months 6 months | 12 months | |
| NYHA class: ( , , , V) | | | |

| eGFR: | | | |
|---|---|---|---|
| Loop diuretics (name,dose): | | | |
| Vital signs | | | |
| | New EF ,method, | , if any : | |
| CV related hospital admission: | ☐ Yes: ☐ WHF ☐ ACS ☐ Arrhythmia S | ☐ Yes: ☐ WHF ☐ ACS ☐ Arrhythmia S | ☐ Yes: ☐ WHF ☐ ACS ☐ Arrhythmias ☐ Others |
| | □ Others | □ Others | 12 months |
| | T | | T |
| | No 3 months 6 months | No | |
| Labs: | | | |
| Meds: | | | |